CLINICAL TRIAL: NCT00743665
Title: Quality of Life And Psychological Symptoms In Children With Cyclic Vomiting Syndrome
Brief Title: Quality of Life And Psychological Symptoms In Children With Cyclic Vomiting Syndrome (CVS)
Status: Completed | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Children's Hospital and Health System Foundation, Wisconsin (Other)
Responsible Party: Principal Investigator, B Li, Professor, Medical College of Wisconsin
Other Study IDs: 07/130; GC 463
Record Dates: First submitted 2008-07-31; First posted 2008-08-29 (Estimated); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Vomiting Syndrome
Keywords: Youth; consensus; criteria; CVS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary aim of this study is to characterize the quality of life of youth with Cyclic Vomiting Syndrome (CVS) as well as the strategies they use to cope with stress, their strengths and vulnerabilities, and to assess symptoms of depression and anxiety in these at risk youth. The impact of CVS on the child's parent and family will also be assessed.

A second aim is to evaluate the associations among coping strategies, personal strengths and vulnerabilities and the frequency and intensity of CVS attacks to determine if particular coping styles and personal characteristics are associated illness severity, psychiatric co-morbidity and quality of life

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CVS

Exclusion Criteria:

* Children and parents who are not English speaking
* Youth with significant developmental delay, mental retardation, psychotic symptoms, or other significant mental impairments and those with other major medical disorders such as IDDM, congenital heart disease, cystic fibrosis, etc.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Youth who meet consensus criteria for CVS as determined by Dr. B. Li and their parents will be recruited from those being seen in the weekly outpatient CVS clinic at Children's Hospital of Wisconsin
Sampling Method: Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2007-06; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sally E Tarbell, PhD, Principal Investigator — Children's Hospital and Health System Foundation, Wisconsin